CLINICAL TRIAL: NCT01249417
Title: A Phase III, Multicentre, Double Blind, Prospective, Randomised, Placebo Controlled Study Assessing the Efficacy and Safety of DYSPORT® Used in the Treatment of Lower Limb Spasticity in Children With Dynamic Equinus Foot Deformity Due to Cerebral Palsy
Brief Title: Dysport® Pediatric Lower Limb Spasticity Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-55-52120-141; 2009-017709-12 (EudraCT Number)
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy; Muscle Spasticity; Children
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dysport 10 U/Kg (Experimental): 10 U/Kg per lower limb. Either one or both lower limbs can be treated. Total volume injected, 2ml per leg.
  Interventions: Biological: Botulinum toxin type A
- Dysport 15 U/Kg (Experimental): 15 U/Kg per lower limb. Either one or both lower limbs can be treated. Total volume injected, 2ml per leg.
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): Total volume to be injected per lower limb - 2ml. Either one or both lower limbs can be treated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — I.M. (in the muscle) injection on day 1 of a single treatment cycle.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport 10 U/Kg; Dysport 15 U/Kg
Drug: Placebo — I.M. injection on day 1 of a single treatment cycle.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine whether Dysport® is effective in the treatment of increased stiffness of the calf muscles and to evaluate the safety of this treatment in children with Cerebral Palsy. In addition this study will also check whether Dysport® can lessen the pain caused by spasticity and improve the child's wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 17 years with cerebral palsy
* Equinus foot position
* Ambulatory
* Intensity of muscle tone equal to or greater than 2 in affected lower limb, as measured on the Modified Ashworth Scale

Exclusion Criteria:

* Fixed contracture
* Previous phenol, alcohol injection or surgical intervention
* Other neurological / neuromuscular disorder
* Severe athetoid or dystonic movements

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (29):
- United States (8):
  - The Children's Hospital, Aurora, Colorado
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Gillette Children's Speciality Healthcare, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriner's Hospital for Children, Portland, Oregon
  - Texas Scottish Rite - Hospital for Children, Dallas, Texas
- Chile (3):
  - Club De Leones Cruz Del Sur Rehabilitation Corporation, Punta Arenas, Punta Arenas
  - Dr Roberto Del Rio Hospital, Santiago
  - Neurorehabilitation Laboratory, Pontifical Catholic University, Santiago
- CHU Jean Minjoz, Besançon, France
- Mexico (4):
  - Hospital San José Celaya, Celaya
  - Centro de Rehabilitacion Infantil, Mexico City
  - Centro de Rehabilitacion Integral de Queretaro (CRIQ), Querétaro
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
- Poland (4):
  - Non-public Healthcare Unit at the Association for Disabled People KROK PO KROKU, Gdansk
  - B i L- Specjalistyczne Centrum Medyczne, Lodz
  - Non-public Healthcare Unit - Grunwaldzka Clinic, Poznan
  - Non-public Healthcare Unit Mazovian Neurorehabilitatio, Wiązowna
- Turkey (Türkiye) (9):
  - Ghulane Military Medical Academy and School of Medicine, Ankara
  - Ibn-i-Sina Hospital, Ankara
  - Yildirim Beyazit Training and Research Hospital, Ankara
  - GATA Haydarpasa Training Hospital, Istanbul
  - Istanbul Fizik Tedavi Rehabilitasyon Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul Fizik Tedavi Rehabilitasyon, Istanbul
  - Istanbul University Medical School, Istanbul
  - Dokuz Eylül University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, İzmit

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each centre that participated in the study was expected to randomise between five and 25 subjects. It was planned to have at least two participating centres per country.
Pre-assignment Details: Screening details:
  A total of 241 subjects were randomised to the study. The safety population included 239 subjects who were treated. Out of the 239 treated subjects, 4 subjects were excluded from the Intent-to-Treat (ITT) population because no MAS score was obtained at the baseline visit and/or at Week 4.
Groups:
- Dysport 10 U/Kg: 10 U/Kg per lower limb. Either one or both lower limbs can be treated. Total volume injected, 2ml per leg.
  Botulinum type A toxin (Dysport®): I.M. (in the muscle) injection on day 1 of a single treatment cycle.
- Dysport 15 U/Kg: 15 U/Kg per lower limb. Either one or both lower limbs can be treated. Total volume injected, 2ml per leg.
  Botulinum type A toxin (Dysport®): I.M. (in the muscle) injection on day 1 of a single treatment cycle.
Period: Randomised Population
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Started | 80 | 80 | 81
Treated (Constitutes the safety population.) | 80 | 80 | 79
Completed | 79 | 79 | 77
Not Completed | 1 | 1 | 4
Not completed — Study treatment not received | 0 | 0 | 2
Not completed — No MAS score at baseline and/or Week 4 | 1 | 1 | 2
Period: Treatment Phase - ITT Population
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Started | 79 | 79 | 77
Completed | 78 | 75 | 73
Not Completed | 1 | 4 | 4
Not completed — Other | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristic values were based on the ITT population, defined as all randomised subjects who received at least one injection of study treatment and who had a MAS score in the GSC assessed both at baseline and at Week 4.
Groups:
- Dysport 10 U/Kg: Dysport 10 U/Kg intramuscular injection on either one or both lower limbs (2 ml per leg), single treatment.
- Dysport 15 U/Kg: Dysport 15 U/Kg intramuscular injection on either one or both lower limbs (2 ml per leg), single treatment.
- Placebo: Placebo intramuscular injection on either one or both lower limbs (2 ml per leg), single treatment.
- Total: Total of all reporting groups
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo | Total
Number analyzed (Participants) | 79 | 79 | 77 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (3.3) | 5.7 (3.2) | 5.9 (3.5) | 5.9 (3.3)
Age, Customized [Number; unit: participants]
  Children (2-9 years) | 67 | 67 | 65 | 199
  Children (10-17 years) | 12 | 12 | 12 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 48 | 141
  Male | 34 | 31 | 29 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 20 | 62
  Not Hispanic or Latino | 58 | 58 | 57 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 2 | 0 | 5 | 7
  Caucasian/White | 57 | 60 | 55 | 172
  American Indian/Alaskan Native | 1 | 0 | 0 | 1
  Multiple | 19 | 19 | 17 | 55
Botulinum toxin Status [Number; unit: participants]
  Naive | 40 | 41 | 41 | 122
  Non-naive | 39 | 38 | 36 | 113
Number of legs being treated [Number; unit: participants]
  1 Leg injected | 42 | 50 | 47 | 139
  2 Legs injected | 37 | 29 | 30 | 96
Gross Motor Function Classification System (GMFCS) [Number; unit: participants] — Participants were staged according to the following GMFCS criteria: level 1 (walks without limitations (best outcome)), level 2 (walks with limitations) and level 3 (walks using a hand held mobility device (worst outcome)). Only participants classified as GMFCS levels 1 to 3 were eligible for entry into the study.
  participants
    GMFCS level 1 | 46 | 45 | 40 | 131
    GMFCS level 2 | 24 | 24 | 30 | 78
    GMFCS level 3 | 9 | 10 | 7 | 26
Height [Mean (Standard Deviation); unit: cm] | 117.1 (20.7) | 111.6 (18.5) | 114.6 (19.7) | 114.4 (19.7)
Weight [Mean (Standard Deviation); unit: kg] | 23.1 (13.4) | 21.1 (10.7) | 22.6 (11.9) | 22.3 (12.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 15.8 (2.9) | 16.1 (2.7) | 16.2 (2.7) | 16.0 (2.8)
Modified Ashworth Scale (MAS) score [Mean (Standard Deviation); unit: units on a scale] — The MAS is a 6-point scale which measures the intensity of muscle tone by measuring the resistance of the muscle to passive lengthening or stretching. The Investigator graded muscle tone in the gastrocnemius-soleus complex (GSC) from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension).
  units on a scale | 3.1 (0.3) | 3.1 (0.3) | 3.2 (0.4) | 3.1 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in MAS Score in the Gastrocnemius-soleus Complex (GSC) at the Ankle Joint of the (Most) Affected Lower Limb
Description: The MAS is a 6-point scale which measures the intensity of muscle tone by measuring the resistance of the muscle to passive lengthening or stretching. Investigator will grade muscle tone in the GSC from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension).
Time Frame: Change from baseline to Week 4
Population: ITT population, defined as all randomised subjects who received at least one injection of study treatment and who had a MAS score in the GSC assessed both at baseline and at Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Number analyzed (Participants) | 79 | 79 | 77
units on a scale | -0.86 [-1.07 to -0.65] | -0.97 [-1.18 to -0.76] | -0.48 [-0.69 to -0.27]
Statistical Analysis 1: Comparison: Dysport 10 U/Kg vs Placebo; LS means for each treatment group and treatment comparisons, as well as the p-values were obtained from an ANCOVA on the change from baseline with treatment, baseline MAS score, age range at baseline, BTX status at baseline and centre as covariates; Test type: Superiority or Other; p = 0.0029, ANCOVA; Difference in LS means = -0.38, 95% CI 2-sided [-0.64 to -0.13]
Statistical Analysis 2: Comparison: Dysport 15 U/Kg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference in LS means = -0.49, 95% CI 2-sided [-0.75 to -0.23]

2. Secondary Outcome: Physician's Global Assessment (PGA) of the Treatment Response.
Description: PGA Scale of the Treatment Response: Global assessment of treatment response assessed by asking the Investigator the following question: "how would you rate the response to treatment in the subject's lower limb(s) since the last injection?" Answers will be made on a 9 point rating scale (-4: markedly worse, -3: much worse, -2: worse, -1: slightly worse, 0: no change, +1: slightly improved, +2: improved, +3: much improved, +4: markedly improved).
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Number analyzed (Participants) | 79 | 79 | 77
units on a scale | 1.54 [1.28 to 1.81] | 1.5 [1.23 to 1.77] | 0.73 [0.46 to 0.99]
Statistical Analysis 1: Comparison: Dysport 10 U/Kg vs Placebo; LS means for each treatment group and treatment comparisons, as well as the p-values were obtained from an ANOVA on the visit value with treatment, age range at baseline, BTX status at baseline and centre as covariates; Test type: Superiority or Other; p < 0.0001, ANOVA; Difference in LS means = 0.82, 95% CI 2-sided [0.50 to 1.14]
Statistical Analysis 2: Comparison: Dysport 15 U/Kg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Difference in LS means = 0.77, 95% CI 2-sided [0.45 to 1.10]

3. Secondary Outcome: Goal Attainment Scale (GAS) Score
Description: GAS is a functional scale used to measure progress towards individual therapy goals. Individual goals defined for each subject by the physician, and the child's parents (caregiver) where applicable, prior to treatment. Post-baseline, the GAS for each goal rated using a defined scale (-2: Much less than expected outcome, -1: somewhat less than expected outcome, 0: expected outcome, 1: somewhat more than expected outcome, and 2: Much more than expected outcome).
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Number analyzed (Participants) | 79 | 79 | 77
units on a scale | 51.53 [49.05 to 54.01] | 50.86 [48.36 to 53.36] | 46.21 [43.7 to 48.72]
Statistical Analysis 1: Comparison: Dysport 10 U/Kg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0006, ANOVA; Difference in LS means = 5.32, 95% CI 2-sided [2.31 to 8.32]
Statistical Analysis 2: Comparison: Dysport 15 U/Kg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0031, ANOVA; LS mean difference = 4.65, 95% CI 2-sided [1.59 to 7.71]

ADVERSE EVENTS:
Time Frame: Up to Week 28 of follow-up
Description: The safety population, defined as all randomised subjects who received at least one injection of study treatment, was used for the analysis of adverse events (AEs).
Arm/Group | Dysport 10 U/Kg | Dysport 15 U/Kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/80 | 4/79
Other Adverse Events (participants affected / at risk) | 51/80 | 51/80 | 42/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 10 U/Kg (N=80) | Dysport 15 U/Kg (N=80) | Placebo (N=79)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 10 U/Kg (N=80) | Dysport 15 U/Kg (N=80) | Placebo (N=79)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (6) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (3) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 8 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (3) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 13 (15) | 10 (11)
Nasopharyngitis (Infections and infestations) | 10 (13) | 9 (10) | 4 (8)
Influenza (Infections and infestations) | 5 (6) | 6 (9) | 6 (7)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (4) | 2 (2)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 6 (7) | 1 (1) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (2) | 4 (5)
Varicella (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No